CLINICAL TRIAL: NCT03634540
Title: A Phase 2 Trial of PT2977 in Combination With Cabozantinib in Patients With Advanced Clear Cell Renal Cell Carcinoma
Brief Title: A Trial of Belzutifan (PT2977, MK-6482) in Combination With Cabozantinib in Patients With Clear Cell Renal Cell Carcinoma (ccRCC) (MK-6482-003)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peloton Therapeutics, Inc., a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6482-003; PT2977-201 (Other: Peloton); MK-6482-003 (Other: MSD)
Record Dates: First submitted 2018-08-03; First posted 2018-08-16 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Renal Cell Carcinoma (RCC); Clear Cell Renal Cell Carcinoma (ccRCC); Kidney Cancer; Renal Cancer; Renal Cell Carcinoma; Renal Cell Cancer Metastatic; Renal Cell Carcinoma Recurrent; Renal Cell Cancer, Recurrent; Kidney
Keywords: hypoxia-inducible factor (HIF); hypoxia-inducible factor 2 alpha (HIF-2α, HIF-2 alpha)
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms; Recurrence | interventions — belzutifan; cabozantinib

STUDY DESIGN:
Intervention Model Description: Belzutifan in combination with cabozantinib administered orally once daily
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Belzutifan + Cabozantinib: Treatment Naïve (Cohort 1) (Experimental): Naïve participants will receive 120 mg belzutifan and 60 mg cabozantinib orally once daily (QD) at the same time.
  Interventions: Drug: Belzutifan; Drug: Cabozantinib
- Belzutifan + Cabozantinib: Prior Immunotherapy (Cohort 2) (Experimental): Participants who have received prior immunotherapy will receive 120 mg belzutifan and 60 mg cabozantinib orally QD at the same time.
  Interventions: Drug: Belzutifan; Drug: Cabozantinib

INTERVENTIONS:
Drug: Belzutifan — Belzutifan tablets administered orally.
  Other Names: PT2977, MK-6482; WELIREG™
Drug: Cabozantinib — Cabozantinib tablets administered orally.
  Other Names: CABOMETYX®

SUMMARY:
This is an open-label Phase 2 study which will evaluate the efficacy and safety of belzutifan in combination with cabozantinib in participants with advanced ccRCC. Belzutifan and cabozantinib will be administered orally once daily.

ELIGIBILITY:
Inclusion Criteria:

* Has locally advanced or metastatic RCC with predominantly clear cell subtype
* Has at least one measurable lesion as defined by RECIST version 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Has adequate organ function defined as follows:

  * Absolute neutrophil count ≥ 1,000/µL, hemoglobin level ≥ 10 g/dL and platelet count ≥ 100,000/µL without transfusion or growth factor support within 2 weeks prior to obtaining the hematology values at screening;
  * Serum creatinine level ≤ 2.0 × upper limit of normal (ULN)
  * Transaminase levels (AST/ALT) ≤ 3.0 × upper limit of normal (ULN); total bilirubin (TBILI) ≤ 1.5 mg/dL in the absence of Gilbert's disease *Cohort 1: Participants must not have received prior systemic therapy for advanced or metastatic ccRCC
* Cohort 2: Participants must have received prior immunotherapy and no more than two prior treatments for advanced or metastatic ccRCC

Exclusion Criteria:

* Has received prior treatment with belzutifan or other HIF2α inhibitors
* Has received prior treatment with cabozantinib
* Has had radiation therapy for bone metastases within two weeks of starting study drug
* Has a history of untreated brain metastases or history of leptomeningeal disease or spinal cord compression
* Has failed to recover from the reversible effects of prior anticancer therapy
* Has uncontrolled or poorly controlled hypertension
* Is receiving anticoagulant therapy
* Has had any major cardiovascular event within 6 months prior to study drug administration
* Has any other clinically significant cardiac, respiratory, or other medical or psychiatric condition that might interfere with participation in the trial or interfere with the interpretation of trial results
* Has had major surgery within 3 months before first study drug administration
* Has an active infection requiring systemic treatment
* Is participating in another therapeutic clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2018-09-27 (Actual); Primary Completion 2027-02-26 (Estimated); Study Completion 2027-02-26 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Up to approximately 2 years
  ORR is defined as the percentage of participants with a best confirmed response of Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions) as determined by the investigator using Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1).

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Up to approximately 2 years
  PFS is defined as the interval from the start of study treatment until the earlier of the first documentation of disease progression determined by RECIST 1.1 or death from any cause.
Duration of Response (DOR) | Up to approximately 2 years
  DOR is defined as the interval from the first documentation of response, as determined by RECIST 1.1, to the earlier of the first documentation of disease progression or death from any cause, and calculated for participants with a best confirmed response of CR (disappearance of all target lesions) or PR (≥30% decrease in the sum of diameters of target lesions).
Time to Response (TTR) | Up to approximately 2 years
  TTR is defined as the interval from the start of study treatment to the first documentation of a response, as determined by RECIST 1.1, and calculated for participants with a best confirmed response of CR or PR.
Overall Survival (OS) | Up to approximately 2 years
  OS is defined as the interval from the start of treatment to the death of the participant from any cause.
Number of participants experiencing an Adverse Event (AE) | Up to approximately 2 years
  An AE is defined as any untoward medical occurrence in a participant regardless of its causal relationship to study treatment. An AE can be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of the study drug, whether or not it is considered to be study drug related. Included in this definition are any newly occurring events and any previous condition that has increased in severity or frequency since the administration of study drug.
Number of participants discontinuing study treatment due to an Adverse Event (AE) | Up to approximately 2 years
  An AE is defined as any untoward medical occurrence in a participant regardless of its causal relationship to study treatment. An AE can be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of the study drug, whether or not it is considered to be study drug related. Included in this definition are any newly occurring events and any previous condition that has increased in severity or frequency since the administration of study drug.
Belzutifan Plasma Concentration | Weeks 1 and 4: pre-dose, 2 and 6 hours post-dose
  Blood samples for the determination of belzutifan concentration will be collected at pre-specified timepoints before and after treatment administration.
Belzutifan Metabolite Plasma Concentration | Weeks 1 and 4: pre-dose, 2 and 6 hours post-dose
  Blood samples for the determination of belzutifan metabolite concentration will be collected at pre-specified timepoints before and after treatment administration.
Cabozantinib Plasma Concentration | Weeks 1 and 4: pre-dose, 2 and 6 hours post-dose
  Blood samples for the determination of cabozantinib concentration will be collected at pre-specified timepoints before and after treatment administration.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (10):
- United States (10):
  - USC Norris Comprehensive Cancer Center ( Site 0060), Los Angeles, California
  - Cedars Sinai Medical Center Samuel Oschin Comp. Cancer Institute ( Site 0003), Los Angeles, California
  - Sylvester Comprehensive Cancer Center ( Site 0023), Miami, Florida
  - Dana Farber Cancer Center ( Site 0006), Boston, Massachusetts
  - Karmanos Cancer Institute ( Site 0033), Detroit, Michigan
  - Tennessee Oncology, PLLC ( Site 0024), Chattanooga, Tennessee
  - Tennessee Oncology, PLLC ( Site 0001), Nashville, Tennessee
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center ( Site 0010), Dallas, Texas
  - Swedish Cancer Institute ( Site 0018), Seattle, Washington
  - Seattle Cancer Care Alliance/Univ of Washington Medical Center ( Site 0035), Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Choueiri TK, McDermott DF, Merchan J, Bauer TM, Figlin R, Heath EI, Michaelson MD, Arrowsmith E, D'Souza A, Zhao S, Roy A, Perini R, Vickery D, Tykodi SS. Belzutifan plus cabozantinib for patients with advanced clear cell renal cell carcinoma previously treated with immunotherapy: an open-label, single-arm, phase 2 study. Lancet Oncol. 2023 May;24(5):553-562. doi: 10.1016/S1470-2045(23)00097-9. Epub 2023 Mar 31. PMID 37011650
- [Derived] Choueiri TK, Merchan JR, Figlin R, McDermott DF, Arrowsmith E, Michaelson MD, Tykodi SS, Heath EI, Spigel DR, D'Souza A, Kassalow L, Perini RF, Vickery D, Bauer TM. Belzutifan plus cabozantinib as first-line treatment for patients with advanced clear-cell renal cell carcinoma (LITESPARK-003): an open-label, single-arm, phase 2 study. Lancet Oncol. 2025 Jan;26(1):64-73. doi: 10.1016/S1470-2045(24)00649-1. PMID 39756444
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com